CLINICAL TRIAL: NCT05510180
Title: Cardiovascular Disease Risk Profile in Children With Hypertrophic Cardiomyopathy
Brief Title: CVD Risk Profile in Children With HCM
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00083230
Record Dates: First submitted 2019-03-05; First posted 2022-08-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertrophic cardiomyopathy is a disease of the heart muscle that causes the heart to become thicker and this thickness places children at risk of heart rhythm problems, heart failure and sudden death.To decrease the risk of sudden death, health care providers generally counsel that the patient should stop all intense physical activity. While this recommendation may decrease the risk of sudden death it is unclear what the long term impact of reduced physical activity is on cardiovascular health in children with HCM.

Cardiovascular (CV) disease is a disease of the heart and blood vessels and is the cause of heart attacks in adults. There are many risk factors for the development of CV disease including genetics, medical conditions and lifestyle choices. While some studies in adults suggest that patients with HCM are at higher risk of poor cardiovascular health, this has not yet been assessed in children. Although, CV disease is generally thought of to be a disease of adults, there is a lot of information that suggests the development of CV disease starts early in life and therefore by promoting heart healthy lifestyles in children, it is possible that these children will becomes healthier adults.

The goal of this project is to assess risk factors for CV disease in a population of children with HCM at the two largest pediatric cardiac programs in Canada. This assessment will be to look at factors we can measure (e.g., weight, cholesterol levels) and patients' and families' perceptions of what it means to be heart healthy. It is hoped that through this project risk factors for heart disease, and poor "heart healthy" lifestyles choices, will be identified in order to develop strategies to decrease these risk factors in patients with HCM. With a better understanding of the families' perceptions of heart healthy behaviours, educational tools and resources for cardiovascular health promotion in patients with HCM can be developed.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is an inherited cardiomyopathy with the hallmark feature of left ventricular hypertrophy primarily involving the ventricular septum. It is associated with an increased risk of arrhythmias and sudden cardiac death (SC) [Maron et al., 2016]. It is the most common genetic heart disease, with a prevalence of up to 1 in 200 in the general population.

It is widely acknowledged that regular physical activity is important for long-term CV health in the general population. Childhood obesity is on the rise in the general population and physicians may be compounding the risk in children with HCM due to the activity restrictions imposed on them. Given the significant emphasis placed on what physical activities patients with HCM should avoid, physicians may not be effectively communicating the importance of maintaining a heart healthy lifestyle, including the importance of regular physical activity, on long-term CV health. This theory could explain the high levels of inactivity and obesity seen in the adult population of individuals with HCM, which have important consequences on long-term health and well-being.

Little research has been done to examine the other markers of CV health in the adult population. In addition, there have not been any studies evaluating the CV disease risk profile of children and adolescents with HCM and whether the phenomenon seen in the adult population is also seen in pediatric patients. This study will fill an important gap which will allow for the development of safe interventions in this unique patient population focused on promoting life-long CV health.

The primary aims of the study are:

1. To describe the CV disease risk behaviors and CV disease risk profile of children with HCM.
2. To determine if children with HCM are at greater risk for acquired CV disease compared to the general population.

The secondary aim of the study are:

1. To identify barriers to a heart healthy lifestyle.
2. To identify both the children's and families' perception of a heart healthy lifestyle.

This study will employ multiple methods. The quantitative component will be a prospective cross-sectional study undertaken at two centers in Canada with a dedicated Heart Function and Cardiomyopathy Department. The quantitative component will be a prospective cross-sectional study undertaken at across pediatric cardiac centers in Canada who look after children with HCM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 10 and 19 years of age meeting the diagnostic criteria for primary hypertrophic cardiomyopathy set in the American Heart Association guideline and their families will be included.
2. Parents and/or guardians of children 10-19 years of age with hypertrophic cardiomyopathy.
3. English speaking -

Exclusion Criteria:

1. Secondary hypertrophic cardiomyopathy
2. Structural congenital heart defects that has the potential to limit physical ability
3. Significant physical disability as identified by the cardiologist that limits physical activity ability (e.g., neuromuscular disease)
4. Significant cognitive disorder or language barrier as identified by the cardiologist that would limit the completion of an English-language survey

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 10 - 19 years of age with primary hypertrophic cardiomyopathy. We are choosing to only include children with HCM as they often are told to not participate in strenuous activities b/c of the risk of sudden death. This patient population also has not been well studied and they often have other co-morbidities that may prevent exercise
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
CV disease risk factors | 2 weeks - Visit 2
  Healthy Hearts School Program Questionnaire
CV disease risk behaviours | 2 weeks - Visit 2
  Healthy Hearts School Program Questionnaire
Acquired CV disease | 2 weeks - Visit 2
  Healthy Hearts School Program Questionnaire

SECONDARY OUTCOMES:
Heart healthy lifestyle barriers | Baseline - Visit 1
  Self-Efficacy for Exercise Scale
Heart healthy lifestyle barriers | Baseline - Visit 1
  PedsQL (Pediatric Quality of Life Inventory and Pediatric Quality of Life Inventory: Cardiac Module)
Child's perception of heart healthy lifestyle | Baseline - Visit 1
  Habitual Activity Estimation Scale (HAES)
Parents' perception of heart healthy lifestyle | Baseline - Visit 1
  Habitual Activity Estimation Scale (HAES)

CONTACTS AND LOCATIONS:
Locations (10):
- Canada (10):
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Université Laval, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No